CLINICAL TRIAL: NCT06276816
Title: Cardiac Denervation Ablation Strategy for Severe Sinus Bradycardia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-LC14
Record Dates: First submitted 2024-01-02; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-11

CONDITIONS: Sinus Bradycardia
Keywords: Sinus Bradycardia; Cardioneuroablation; Sinus Node Dysfunction; Autonomic Nervous System
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective clinical observation and registration study. The investigator aimed to evaluate the efficacy and safety of cardiac denervation ablation as a treatment strategy for severe sinus bradycardia.

DETAILED DESCRIPTION:
Severe sinus bradycardia (SSB) is a common clinical condition that can lead to symptoms such as dizziness, fainting, and even cardiac arrest, posing a serious threat to patients' health and life. The causes of SSB vary: in elderly patients, SSB is often caused by ischemia and degenerative changes in the sinoatrial node, while in younger patients, it is often due to abnormal elevation of vagal nerve tone resulting in slowed heart rate and weakened myocardial contractility. Although implanting a pacemaker can effectively alleviate SSB bradycardia, the incidence of pacemaker electrode-related complications (such as electrode displacement, insulation layer rupture, lead infection, and fracture) is not low. Moreover, the impact of pacemaker implantation on patients' quality of life and the economic burden of regular pacemaker battery replacement impose significant psychological and financial burdens on patients, especially young patients. Clearly, for young SSB patients, if the abnormally elevated vagal nerve tone can be continuously reduced, it would be more effective in treating bradycardia and avoiding pacemaker implantation, which has significant social and economic value.

The investigators has pioneered the technique of cardiac denervation ablation, which can modulate the autonomic nervous tone of the heart and is used to treat autonomic nervous system-related diseases. In a preliminary exploratory study involving 6 SSB patients, investigators found that cardiac denervation ablation for SSB can reduce vagal nerve tone, increase sinus heart rate, and effectively alleviate bradycardia symptoms, thus avoiding the need for pacemaker implantation.

Therefore, based on the preliminary work, this project aims to conduct a prospective observational study and establish a registry. SSB patients who meet the indications for pacemaker implantation will be selected to evaluate the efficacy and safety of cardiac denervation ablation for SSB, its impact on quality of life, and the effectiveness of avoiding pacemaker implantation. The project will establish standardized surgical strategies and protocols for cardiac denervation ablation for SSB, summarize experiences, and lay the foundation for the clinical promotion and guideline revision of catheter ablation for SSB.

ELIGIBILITY:
Inclusion Criteria:

1. Sinus bradycardia and pacemaker implantation indication: long interval with mean heart rate <45 bpm or 3s recorded within 6 months before inclusion;
2. Negative atropine test: sinus heart rate> 90bpm after atropine injection
3. SSB related symptoms: dizziness, palpitations, fatigue, amaurosis, syncope, etc.
4. Age ≥18 and <60 years old;
5. The patient has agreed to participate in this trial and has signed the informed consent form.

Exclusion Criteria:

1. Previous history of atrial arrhythmia ablation or surgical procedure;
2. Structural heart disease, chronic liver and kidney dysfunction, diabetes mellitus, neurological diseases.;
3. Drug-related SSB;
4. presence of left atrial thrombus;
5. Pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: SSB patients undergoing cardiac denervation ablation
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with postoperative recurrence of bradycardia symptoms | 12 months after ablation procedure
  Symptoms such as chest tightness, suffocation, amaurosis, syncope with cardiac arrest with mean heart rate <45bpm or ≥3s on 12-lead ECG or Holter

SECONDARY OUTCOMES:
The result of the atropine test | 12 months after ablation procedure
  A negative response was defined as a 25% increase in sinus heart rate or an increase in sinus rhythm to 90 bpm after atropine injection.
Changes in quality of life measured by Medical Outcomes Study 36- Item Short Form Health Survey (SF-36) | 3, 6, 12 months after ablation procedure
  Patients' quality of life was assessed by Medical Outcomes Study 36- Item Short Form Health Survey (SF-36). The scale contains 36 items in 9 categories of physical functioning, role-physica, bodily pain, general health, vitality, social functioning, role-emotional, mental health and reported health transition. Subjects' scores ranged from 0 to 900, with higher scores representing better quality of life.
Changes in quality of life measured by EuroQol Five Dimensions Questionnaire Visual Analogue Scale (EQ VAS) | 3, 6, 12 months after ablation procedure
  Patients' quality of life was assessed by EuroQol Five Dimensions Questionnaire Visual Analogue Scale (EQ VAS). Subjects' scores ranged from 0 to 100, with higher scores representing better quality of life.
Changes in minmum heart rate | 3, 6, 12 months after ablation procedure
  Comparison of postoperative versus baseline minimum heart rate using a 24-hour holter. The device provided to patients prior to discharge or at outpatient visits will be used for this assessment.
Changes in mean heart rate | 3, 6, 12 months after ablation procedure
  Comparison of postoperative versus baseline mean heart rate using a 24-hour holter. The device provided to patients prior to discharge or at outpatient visits will be used for this assessment.
Changes in deceleration capacity | 3, 6, 12 months after ablation procedure
  Comparison of postoperative versus baseline deceleration capacity (DC) using a 24-hour holter. Higher DC suggest higher vagal activity. The device provided to patients prior to discharge or at outpatient visits will be used for this assessment.

CONTACTS AND LOCATIONS:
Overall Officials: yan Yao, PhD, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases
Locations (1):
- 1Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

REFERENCES:
- [Result] Shen WK, Sheldon RS, Benditt DG, Cohen MI, Forman DE, Goldberger ZD, Grubb BP, Hamdan MH, Krahn AD, Link MS, Olshansky B, Raj SR, Sandhu RK, Sorajja D, Sun BC, Yancy CW. 2017 ACC/AHA/HRS Guideline for the Evaluation and Management of Patients With Syncope: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2017 Aug 1;136(5):e60-e122. doi: 10.1161/CIR.0000000000000499. Epub 2017 Mar 9. No abstract available. PMID 28280231
- [Result] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Result] Sun W, Zheng L, Qiao Y, Shi R, Hou B, Wu L, Guo J, Zhang S, Yao Y. Catheter Ablation as a Treatment for Vasovagal Syncope: Long-Term Outcome of Endocardial Autonomic Modification of the Left Atrium. J Am Heart Assoc. 2016 Jul 8;5(7):e003471. doi: 10.1161/JAHA.116.003471. PMID 27402231
- [Result] Hu F, Zheng L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Right anterior ganglionated plexus: The primary target of cardioneuroablation? Heart Rhythm. 2019 Oct;16(10):1545-1551. doi: 10.1016/j.hrthm.2019.07.018. Epub 2019 Jul 19. PMID 31330187
- [Result] Hu F, Zheng L, Liu S, Shen L, Liang E, Liu L, Wu L, Ding L, Yao Y. The impacts of the ganglionated plexus ablation sequence on the vagal response, heart rate, and blood pressure during cardioneuroablation. Auton Neurosci. 2021 Jul;233:102812. doi: 10.1016/j.autneu.2021.102812. Epub 2021 Apr 20. PMID 33940549
- [Result] Hu F, Zheng L, Liu S, Shen L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Avoidance of Vagal Response During Circumferential Pulmonary Vein Isolation: Effect of Initiating Isolation From Right Anterior Ganglionated Plexi. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007811. doi: 10.1161/CIRCEP.119.007811. Epub 2019 Nov 25. PMID 31760820
- [Result] Tu B, Wu L, Hu F, Fan S, Liu S, Liu L, Ding L, Zheng L, Yao Y. Cardiac deceleration capacity as an indicator for cardioneuroablation in patients with refractory vasovagal syncope. Heart Rhythm. 2022 Apr;19(4):562-569. doi: 10.1016/j.hrthm.2021.12.007. Epub 2021 Dec 9. PMID 34896621
- [Result] Zheng L, Sun W, Qiao Y, Hou B, Guo J, Killu A, Yao Y. Symptomatic Premature Ventricular Contractions in Vasovagal Syncope Patients: Autonomic Modulation and Catheter Ablation. Front Physiol. 2021 May 3;12:653225. doi: 10.3389/fphys.2021.653225. eCollection 2021. PMID 34012407
- [Result] Stavrakis S, Scherlag BJ, Po SS. Autonomic modulation: an emerging paradigm for the treatment of cardiovascular diseases. Circ Arrhythm Electrophysiol. 2012 Apr;5(2):247-8. doi: 10.1161/CIRCEP.112.972307. No abstract available. PMID 22511657
- [Result] Zhao L, Jiang W, Zhou L, Wang Y, Zhang X, Wu S, Xu K, Liu X. Atrial autonomic denervation for the treatment of long-standing symptomatic sinus bradycardia in non-elderly patients. J Interv Card Electrophysiol. 2015 Aug;43(2):151-9. doi: 10.1007/s10840-015-9981-8. Epub 2015 Feb 19. PMID 25693516
- [Result] Qin M, Zhang Y, Liu X, Jiang WF, Wu SH, Po S. Atrial Ganglionated Plexus Modification: A Novel Approach to Treat Symptomatic Sinus Bradycardia. JACC Clin Electrophysiol. 2017 Sep;3(9):950-959. doi: 10.1016/j.jacep.2017.01.022. Epub 2017 Apr 26. PMID 29759719
- [Result] Debruyne P, Rossenbacker T, Collienne C, Roosen J, Ector B, Janssens L, Charlier F, Vankelecom B, Dewilde W, Wijns W. Unifocal Right-Sided Ablation Treatment for Neurally Mediated Syncope and Functional Sinus Node Dysfunction Under Computed Tomographic Guidance. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006604. doi: 10.1161/CIRCEP.118.006604. PMID 30354289
- [Result] Debruyne P, Rossenbacker T, Janssens L, Collienne C, Ector J, Haemers P, le Polain de Waroux JB, Bazelmans C, Boussy T, Wijns W. Durable Physiological Changes and Decreased Syncope Burden 12 Months After Unifocal Right-Sided Ablation Under Computed Tomographic Guidance in Patients With Neurally Mediated Syncope or Functional Sinus Node Dysfunction. Circ Arrhythm Electrophysiol. 2021 Jun;14(6):e009747. doi: 10.1161/CIRCEP.120.009747. Epub 2021 May 17. PMID 33999698